CLINICAL TRIAL: NCT00279006
Title: Adhesiveness of Coronary Drug-Eluting Stents to the Delivery Balloon-Catheter: A Randomized Comparison
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Foundation for Cardiovascular Research, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK-12006
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2006-01

CONDITIONS: Coronary Artery Disease
Keywords: DES (drug eluting stents); CAD (cornary artery disease); stent retrieval
MeSH Terms: conditions — Coronary Artery Disease; Dysequilibrium syndrome | interventions — Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention

SUMMARY:
This study will evaluate the 3 drug-eluting stents presently marketed for intervention in the coronary artery with respect to the complications that may occur in case it becomes necessary to retract the stent during the intervention. It has been noted that stents carrying a drug for local application may be more difficult to retract than the more smooth bare metal stents.

DETAILED DESCRIPTION:
Patients in whom DES implantation is planned will be randomized to one of the 3 commercially available stents (i.e., Cypher, Taxus-Liberté, Endeavor).

Sealed envelopes will be used for randomization purposes. Should additional stents be required in the same patient for the same or other lesions, another stent of the same type of stents will be implanted.

The following assessments will be made:

* Unblinded subjective operator assessment based on a questionnaire. The questionnaire will include questions on problems encountered during stent-balloon retrieval, special maneuvers performed (e.g., retrieval of the catheter during device removal, and possible complications associated with device retrieval).
* Blinded measurements of following parameters:

  1. Minimal and maximal distance between the tip of the guiding catheter and the proximal stent end during stent-balloon retrieval.
  2. Minimal and maximal distance between the tip of the guidewire and the distal portion of the stent during stent-balloon retrieval.
  3. To do so the retrieval of the stent-balloon will be documented on ciné-angiography. The measurements will be performed by a qualified technician/physician blinded to the type of device used.
* Clinical endpoints:

  d. In-Hospital mortality, myocardial infarction, or need for unplanned urgent repeat revascularization.

  e. Myocardial infarction defined as creatine kinase MB-isoform [CK-MB] ≥3x upper limit of normal within 24 hours of the procedure or ≥2x upper limit of normal after 24 hours of the procedure in the presence of new ischemic symptoms.
* Target enrollment of 150 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with a planned angiography and percutane coronary intervention
* Age 18 years or above
* Informed consent to PCI and to participation in this trial

Exclusion Criteria:

* Patients who after angiography are deemed not suitable for stent implant (operators discretion)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-01; Study Completion 2007-03

PRIMARY OUTCOMES:
In-Hospital mortality, myocardial infarction, or need for unplanned urgent repeat revascularization.
Myocardial infarction defined as creatine kinase MB-isoform [CK-MB] ≥3x upper limit of normal within 24 hours of the procedure or ≥2x upper limit of normal after 24 hours of the procedure in the presence of new ischemic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Franz R Eberli, MD, Study Director — University Hospital, Zürich